CLINICAL TRIAL: NCT03787472
Title: Clinical Evaluation of Manufacturing Curing Processes for a Reusable Multifocal Optical Design in a Presbyopic Population
Brief Title: Clinical Evaluation of Manufacturing Processes for a Reusable Multifocal Optical Design in a Presbyopic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6317
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Hyperopic subjects that are habitual soft contact lens wearers and have presbyopia will be randomized into one the sequence (Test/Control).
  Interventions: Device: JJV Investigational senofilcon A Multifocal Lens1; Device: JJV Investigational senofilcon A Multifocal Lens2
- Control/Test (Experimental): Hyperopic subjects that are habitual soft contact lens wearers and have presbyopia will be randomized into the sequence (Control/Test).
  Interventions: Device: JJV Investigational senofilcon A Multifocal Lens1; Device: JJV Investigational senofilcon A Multifocal Lens2

INTERVENTIONS:
Device: JJV Investigational senofilcon A Multifocal Lens1 — CONTROL
Device: JJV Investigational senofilcon A Multifocal Lens2 — TEST

SUMMARY:
The clinical study is a randomized-controlled, double-masked, crossover clinical trial with two study treatments to compare two study lens types and the initial performance, in terms of the subjective response after a period of lens dispensing. The study will last approximately 2 to 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be at least 40 years of age and not greater than 70 years of age.
  4. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
  5. The subject's refractive cylinder must be ≤0.75 D in each eye.
  6. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  7. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.
  8. Subjects must own a wearable pair of spectacles if required for their distance vision.
  9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).
  10. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
  6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy cataract surgery, retinal surgery, etc.).
  7. A history of amblyopia, strabismus or binocular vision abnormality.
  8. Any current ocular infection or inflammation.
  9. Any current ocular abnormality that may interfere with contact lens wear.
  10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, systemic steroids.
  11. Use of any ocular medication, with the exception of rewetting drops.
  12. History of herpetic keratitis.
  13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  15. Any known hypersensitivity or allergic reaction to Optifree®Replenish® multipurpose care solution, sodium fluorescein or Eye-Cept® rewetting drop solution.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Maitland Vision Center, Maitland, Florida
  - Advanced Eyecare, Raytown, Missouri
  - Spectrum Eyecare, Jamestown, New York
  - Western Reserve Vision Care, Inc, Beachwood, Ohio
  - ProCare Vision Centers, Granville, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 subjects were enrolled in this study and all 45 subjects were randomly assigned to one of the two lens sequences and completed the study. 3 subjects were excluded from analysis and 42 were included in Per-Protocol Population.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to the Protocol Deviation, 3 subjects were excluded from the analysis population.
Groups:
- Total: All subjects who had successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock.
Arm/Group | Total
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1
  White | 41
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: CLUE Vision
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test: Subjects that wore the Test lens in either the first or second period of the study.
- Control: Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 42 | 42
units on a scale | 52.77 (18.872) | 52.23 (19.54)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — The non-inferiority of the Test lens relative to the Control will be concluded if the lower confidence limit of LSM difference is above the non-inferiority margin -5; Linear Mixed Model; The Kenward and Roger method was used for the calculation of the denominator of degrees of freedom; Least-Square Mean Difference = 0.5, 95% CI 2-sided [-5.5 to 6.6], Standard Error of Mean 2.98 — Mean difference was calculated as Test - Control

2. Secondary Outcome: logMAR Visual Acuity
Description: Binocular visual performance on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated under high luminance and high contrast conditions at three distances:
  Distance (3 meters) was measured using ETDRS (Early Treatment Diabetic Retinopathy Study) charts; Intermediate (64 centimeters) and Near (40 centimeters) were measured using Reduced Guillon-Poling Charts.
  Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR units
Units Other Than Participants: Eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 42 | 42
Number analyzed (Eyes) | 84 | 84
logMAR units
  Distance Standard High Contrast Bright | -0.088 (0.0885) | -0.096 (0.0938)
  Intermediate Standard High Contrast Bright | -0.047 (0.0863) | -0.035 (0.0950)
  Near Standard High Contrast Bright | 0.080 (0.0908) | 0.076 (0.0903)
Statistical Analysis 1: Comparison: Test vs Control; Distance Standard High Contrast Bright; Test type: Non-Inferiority — The non-inferiority of the Test lens relative to the Control will be concluded if the upper confidence limit of LSM difference is below the non-inferiority margin 0.05 logMAR; Linear Mixed Model; Least-Square Mean Difference = 0.008, 95% CI 2-sided [-0.025 to 0.041], Standard Error of Mean 0.0166 — Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Test vs Control; Intermediate Standard High Contrast Bright; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Linear Mixed Model; Least-Square Mean Difference = -0.012, 95% CI 2-sided [-0.043 to 0.019], Standard Error of Mean 0.0155 — Mean difference was calculated as Test - Control
Statistical Analysis 3: Comparison: Test vs Control; Near Standard High Contrast Bright; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Linear Mixed Model; Least-Square Mean Difference = 0.003, 95% CI 2-sided [-0.030 to 0.037], Standard Error of Mean 0.0169 — Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 5 weeks per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03787472/Prot_SAP_000.pdf